CLINICAL TRIAL: NCT00800241
Title: Budesonide/Formoterol for Maintenance and Reliever Therapy: A Medication Use Evaluation Among Persistent Asthma Patients in General Practice in Thailand
Brief Title: Budesonide/Formoterol for Maintenance and Reliever Therapy Among Asthma Patients in Thailand
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Thanu Komolsai, MD, Medical Advisor, AstraZeneca (Thailand) Ltd.
Other Study IDs: NIS-RTH-SYM-2008/1
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Asthma
Keywords: Asthma; Symbicort SMART; Thai patient eligibility; Persistent asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the incidence of misuse, i.e., over-use and under-use, of Budesonide/formoterol for maintenance and reliever therapy in usual-care setting.

ELIGIBILITY:
Inclusion Criteria:

* Established persistent asthma
* Currently treated with Symbicort SMART for 3 months or longer

Exclusion Criteria:

* currently participating or have participated in a study with an investigational compound within the last 30 days
* current diagnosis of chronic obstructive pulmonary disease (COPD)
* smoked more than 10 pack-year

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient aged 12 years or older who established persistent asthma and currently treated with Symbicort SMART for 3 months or longer.
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Estimated)
Dates: Start 2009-05; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Number of budesonide/formoterol use per patient | On the survey date

CONTACTS AND LOCATIONS:
Overall Officials: Bandit Thinkhamrop, PhD., Principal Investigator — Department of Biostatistics and Demography, Faculty of Public Health, Khon Kaen University; Watchara Boonsawat, MD, PhD, Principal Investigator — Department of Medicine, Faculty of Medicine, Khon Kaen University
Locations (14):
- Thailand (14):
  - Research Site, Buriram
  - Research Site, Chanthaburi
  - Research Site, Chiang Mai
  - Research Site, Mahasarakham
  - Research Site, Nakhon Phanom
  - Research Site, Nakhon Srithammarat
  - Research Site, Nakhonpathom
  - Research Site, Phatthalung
  - Research Site, Phitsanulok
  - Research Site, Rayong
  - Research Site, Roi Et
  - Research Site, Samutsakhon
  - Research Site, Surat Thani
  - Research Site, Trang